CLINICAL TRIAL: NCT01003535
Title: Quantification of Cerebral Cholinergic Function in Patients With Parkinson´s Disease by Means of Nuclear Medicine Methods
Brief Title: Quantification of Cerebral Cholinergic Function in Parkinson´s Disease by Means of Nuclear Medicine Methods
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Joerg Spiegel, M.D, Universität des Saarlandes
Other Study IDs: JoergSpiegel1
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Parkinson´s Disease; Acetylcholine; SPECT
Keywords: Parkinson´s disease; Acetylcholine receptors
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- [123I]5-IA-85380 SPECT

SUMMARY:
Parkinson´s disease is based on a Lewy body degeneration of cerebral and extracerebral neurons. This Lewy body degeneration includes cerebral cholinergic neurons besides dopaminergic neurons.

In previous studies the investigators found that some clinical parkinsonian symptoms - primarily hypokinesia and rigidity - significantly correlate with the dopaminergic nigrostriatal degeneration which was quantified by dopamine transporter imaging. In contrast to that, resting or postural parkinsonian tremor does not correlate with the dopaminergic nigrostriatal degeneration. Obviously further cerebral changes - for instance possible changes / degeneration of cerebral cholinergic neurons - contribute to parkinsonian tremor.

In this study the investigators apply cerebral 5-IA-85380-SPECT to quantify the local density of cerebral nicotinergic cholinergic receptors in patients with Parkinson´s disease. The investigators will correlate the results of cerebral 5-IA-85380-SPECT with the clinical parkinsonian main symptoms hypokinesia, rigidity and primarily resting and postural tremor. In particular, it is of interest whether changes of cerebral cholinergic neurons are involved in the generation of parkinsonian tremor.

DETAILED DESCRIPTION:
The protocol of our study - as explained in the following - was approved by the Local Ethics committee (Ethics committee of the medical association of the Saarland, D-66111 Saarbrücken, Germany, file number 201/06) and by the German Federal Agency for Radiation Protection (Bundesamt für Strahlenschutz, D-38201 Salzgitter, Germany, file number Z 5 - 22461/2 2008-207).

Aims of this study:

In this study we measure the density and local distribution of cerebral acetylcholine receptors in patients with Parkinson´s disease (PD) by means of [123I]5-IA-85380 SPECT. [123I]5-IA-85380 SPECT was applied in healthy volunteers (Fujita et al. 2002, Fujita et al. 2003, Ding et al. 2004, Mamede et al. 2004, Obrzut et al. 2005) and PD patients (Fukuyama et al. 2004, Bucerius et al. 2006, Fujita et al. 2006). These numerous previous studies proved that [123I]5-IA-85380 SPECT is a safe and effective method to visualize cerebral acetylcholine receptors.

We intend to correlate the density and distribution of cerebral acetylcholine receptors with the clinical parkinsonian cardinal symptoms tremor, hypokinesia and rigidity. The patients are out-patients who are treated by the Department of Neurology, Saarland University, D-66421 Homburg/Saar, Germany. The nuclear medicine measurement [123I]5-IA-85380 SPECT will be performed in the Department of Nuclear medicine of the University of Würzburg, D-97080 Würzburg, Germany.

This study should answer the following questions:

1. Does the density of acetylcholine receptors in putamen, caudate nucleus, thalamus and pons correlate with the severity of the clinical symptoms hypokinesia, rigidity, resting tremor, postural tremor?
2. Do PD patients with the tremor dominant type, akinetic rigid type and equivalence type differ concerning their accumulation of 5-IA-85380 (=density of acetylcholine receptors) in the putamen, caudate nucleus, thalamus and pons?

Study protocol:

This study will include 25 patients with Parkinson´s disease (PD), Hoehn and Yahr stage 1. 25 patients have to be included ,if a correlation coefficient r = 0.5, an error 1st order = 0.05 and an error 2nd order = 0.20 are assumed. In addition, the number of 25 patients was sufficient in previous studies to obtain significant results. Due to the stochastic risk of radiation-induced long-term side effects (for example neoplasms), which is higher in younger patients, the lower age limit of included patients is determined to 50 years. The upper age limit is 75 years, since vascular cerebral changes increase exponentially in the higher age. The antiparkinsonian medication - except anticholinergic medication - can be continued during the nuclear medicine examination because previous studies excluded any interference between antiparkinsonian medication - except anticholinergic medication - and 5-IA-85380 SPECT.

The severity of the clinical parkinsonian motor symptoms hypokinesia, rigidity, resting tremor and postural tremor are quantified by means of the motor part of the UPDRS (Unified Parkinson´s Disease Rating Scale). The UPDRS is measured in the "Off"-state; "Off"-state means that the medication was interrupted for at least twelve hours. Further the Mini Mental State-Test and DemTect are measured. Healthy controls are not included since there exist norm values in the literature (Fujita et al. 2002, Fujita et al. 2003, Ding et al. 2004, Mamede et al. 2004, Obrzut et al. 2005).

The tracer [123I]5-IA-85380 is produced in the laboratory of radiochemistry and radiopharmacy of the University of Würzburg at the day of examination. This laboratory has the official permission to produce radiotracers. After informed consent by the patient and thyroid gland blocking with perchlorate, the radioactively marked tracer [123I]5-IA-85380 (185 MBq) was given intravenously. Cerebral SPECT imaging was performed 2-3 hours after intravenous injection of the radioactive substance [123I]5-IA-85380. A triple-head gamma camera equipped with low-energy high-resolution collimators was used. Data was acquired in a 128 x 128 matrix covering 120 degrees per camera and head, 50 seconds per view. A total of 120 views was acquired.

Statistical analysis:

The correlation between density of acetylcholine receptors (= uptake of [123I]5-IA-85380) in different brain regions is correlated with the severity of clinical symptoms. The latter was quantified by the items of the UPDRS score.

Correlations were calculated using the Pearson´s correlation coefficient in case of a normally distributed data and Spearman´s correlation coefficient in case of a not normally distributed data.

ELIGIBILITY:
Inclusion Criteria:

* patients with Parkinson´s disease (after the UK Brain Bank criteria)
* Hoehn and Yahr stage 1
* age 50 - 75 years
* non-smokers
* informed consent to participate in the study

Exclusion Criteria:

* pregnant or nursing women
* no adequate contraception in women who are capable of childbearing
* male patients living with fertile women without adequate contraception
* smokers
* actual or past drug or alcohol abuse
* dementia (minimental state test < 25 points)
* psychosis or antipsychotic medication in the last 12 months
* cholinergic or anticholinergic medication
* unstable or severe internal diseases

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson´s disease
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Correlation of density of acetylcholine receptors in distinct brain areas versus the clinical parameters resting tremor, postural tremor, hypokinesia and rigidity in patients with Parkinson´s disease | 1 time

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Spiegel, M.D., Principal Investigator — Department of Neurology, Saarland University, Kirrberger Strasse, D-66421 Homburg/Saar, Germany
Locations (1):
- Department of Neurology, Saarland University, Homburg/Saar, Saarland, Germany

REFERENCES:
- [Background] Bucerius J, Joe AY, Schmaljohann J, Gundisch D, Minnerop M, Biersack HJ, Wullner U, Reinhardt MJ. Feasibility of 2-deoxy-2-[18F]fluoro-D-glucose- A85380-PET for imaging of human cardiac nicotinic acetylcholine receptors in vivo. Clin Res Cardiol. 2006 Feb;95(2):105-9. doi: 10.1007/s00392-006-0342-6. Epub 2006 Jan 19. PMID 16598519
- [Background] Ding YS, Fowler JS, Logan J, Wang GJ, Telang F, Garza V, Biegon A, Pareto D, Rooney W, Shea C, Alexoff D, Volkow ND, Vocci F. 6-[18F]Fluoro-A-85380, a new PET tracer for the nicotinic acetylcholine receptor: studies in the human brain and in vivo demonstration of specific binding in white matter. Synapse. 2004 Sep 1;53(3):184-9. doi: 10.1002/syn.20051. No abstract available. PMID 15236351
- [Background] Fujita M, Seibyl JP, Vaupel DB, Tamagnan G, Early M, Zoghbi SS, Baldwin RM, Horti AG, KoreN AO, Mukhin AG, Khan S, Bozkurt A, Kimes AS, London ED, Innis RB. Whole-body biodistribution, radiation absorbed dose, and brain SPET imaging with [123i]5-i-A-85380 in healthy human subjects. Eur J Nucl Med Mol Imaging. 2002 Feb;29(2):183-90. doi: 10.1007/s00259-001-0695-z. PMID 11926380
- [Background] Fujita M, Ichise M, van Dyck CH, Zoghbi SS, Tamagnan G, Mukhin AG, Bozkurt A, Seneca N, Tipre D, DeNucci CC, Iida H, Vaupel DB, Horti AG, Koren AO, Kimes AS, London ED, Seibyl JP, Baldwin RM, Innis RB. Quantification of nicotinic acetylcholine receptors in human brain using [123I]5-I-A-85380 SPET. Eur J Nucl Med Mol Imaging. 2003 Dec;30(12):1620-9. doi: 10.1007/s00259-003-1320-0. Epub 2003 Oct 2. PMID 14523584
- [Background] Fujita M, Ichise M, Zoghbi SS, Liow JS, Ghose S, Vines DC, Sangare J, Lu JQ, Cropley VL, Iida H, Kim KM, Cohen RM, Bara-Jimenez W, Ravina B, Innis RB. Widespread decrease of nicotinic acetylcholine receptors in Parkinson's disease. Ann Neurol. 2006 Jan;59(1):174-7. doi: 10.1002/ana.20688. PMID 16374823
- [Background] Fukuyama H. Functional brain imaging in Parkinson's disease-overview. J Neurol. 2004 Oct;251 Suppl 7:vII1-3. doi: 10.1007/s00415-004-1702-7. No abstract available. PMID 15505748
- [Background] Mamede M, Ishizu K, Ueda M, Mukai T, Iida Y, Fukuyama H, Saga T, Saji H. Quantification of human nicotinic acetylcholine receptors with 123I-5IA SPECT. J Nucl Med. 2004 Sep;45(9):1458-70. PMID 15347712
- [Background] Obrzut SL, Koren AO, Mandelkern MA, Brody AL, Hoh CK, London ED. Whole-body radiation dosimetry of 2-[18F]Fluoro-A-85380 in human PET imaging studies. Nucl Med Biol. 2005 Nov;32(8):869-74. doi: 10.1016/j.nucmedbio.2005.06.005. PMID 16253812